CLINICAL TRIAL: NCT05262777
Title: A Randomized, Evaluator-blinded, Parallel Group, Comparator-controlled, Multicenter Study to Evaluate the Safety and Effectiveness of GP0112 for Cheek Augmentation and Correction of Midface Contour Deficiencies
Brief Title: Safety and Effectiveness of GP0112 for Cheek Augmentation and Correction of Midface Contour Deficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43N1CA2104
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cheek Wrinkles; Midface Contour Deficiencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP0112 (Experimental): GP0112 Single injection and optional touch up injection and re-treatment with GP0112
  Interventions: Device: GP0112
- Restylane Lyft Lidocaine (Active Comparator): Restylane Lyft Lidocaine Single injection and optional touch up injection and re-treatment with Restylane Lyft Lidocaine
  Interventions: Device: Restylane Lyft Lidocaine

INTERVENTIONS:
Device: GP0112 — Injectable gel
  Arms: GP0112
Device: Restylane Lyft Lidocaine — Injectable gel
  Arms: Restylane Lyft Lidocaine

SUMMARY:
A randomized, evaluator-blinded, parallel group, comparator-controlled, multicenter study to evaluate the safety and effectiveness of GP0112 for cheek augmentation and correction of midface contour deficiencies

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Men and non-pregnant, non-breastfeeding women aged 18 years or older.
3. MMVS grade of 2, 3 or 4 (mild to substantial loss of fullness in the midface area) on each side of the face as assessed by the Blinded Evaluator. The MMVS for each side of the face does not need to be equal, however the difference between the two sides should be limited to 1 grade.
4. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study (e.g., laser or chemical resurfacing, needling, facelift, lifting threads, radiofrequency etc.).
5. Intent to undergo treatment for correction of midface volume deficit.

   Inclusion criteria 6-7 apply to female subjects only
6. If the subject is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at the screening/baseline visit, prior to treatment/injection, and at the end of study visit.
7. Negative UPT for women of childbearing potential at the screening/baseline visit and all injection visits.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins.
2. Known/previous allergy or hypersensitivity to local anesthetics, e.g. lidocaine or other amide-type anesthetics or nerve blocking agents (if intended to be used for that subject).
3. Previous or present severe or multiple allergies manifested by severe reactions, such as anaphylaxis or angioedema, or family history of these conditions.
4. Previous facial surgery (e.g. facial fat removal, facelift and sinus surgery) in or near the treatment area that in the Treating Investigator´s opinion could interfere with the study safety and/or effectiveness assessments.
5. Any previous aesthetic procedures or implants:

   * Previous use of any permanent (non-biodegradable) or semi-permanent (e.g., calcium hydroxylapatite or Poly-L-Lactic acid) facial tissue augmentation therapy, lifting threads, permanent implants or autologous fat in the face regardless of time.
   * Previous HA filler or collagen filler in or near the treatment area within 12 months.
   * Previous botulinum toxin treatment in or near the treatment area within 6 months.
   * Previous energy based aesthetic procedures (e.g. laser, intense pulsed light, radiofrequency and ultrasound) in or near the treatment area within 6 months.
   * Previous mechanical (e.g. dermabrasion, needling) or chemical aesthetic procedures (e.g. chemical peel) in or near the treatment area within 6 months.
   * Previous treatment with cryotherapy in or near the treatment area within 6 months.
6. History of cancer or previous radiation near or on the area to be treated.
7. Presence of any disease or lesions near or on the area to be treated, e.g.,

   * Inflammation, active or chronic infection (e.g., in mouth, dentals, head);
   * Facial psoriasis, eczema, acne, rosacea, perioral dermatitis, herpes simplex or herpes zoster;
   * Scars or deformities;
   * Cancer, or precancerous conditions (e.g. actinic keratosis or actinic cheilitis).
8. Evidence of scar-related disease or delayed healing activity within 1 year prior to the baseline visit, or subjects susceptible to keloid formation, hyperpigmentation or hypertrophic scarring.
9. Presence of tattoo, piercing, beard or facial hair, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
10. Presence of a dental, oral, or facial condition which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment; e.g. has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities. Any planned procedure (e.g. dental implants, tooth extractions, orthodontia) during the study period, that would make the subject unsuitable for inclusion in the opinion of the Investigator.
11. An underlying known disease, a surgical or medical condition that would expose the subject to undue risk, e.g. human immunodeficiency virus (HIV), active hepatitis, autoimmune disease, history of bleeding disorders, connective tissue diseases such as rheumatoid arthritis, systemic lupus erythematosus, polymyositis, dermatomyositis, or scleroderma.
12. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g. aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard multivitamin formulation.
13. Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. immunosuppressive monoclonal antibodies, antiviral treatment for HIV or hepatitis).
14. Treatment with systemic corticosteroids (inhaled corticosteroids are allowed) within 3 months prior to Baseline visit.
15. Use of topical facial corticosteroids or prescription retinoids near or on the area to be treated within 1 month of the Baseline visit or systemic retinoid treatment within 6 months of the Baseline visit, or plan to receive such treatment during participation in the study.
16. Presence of any condition or situation, which in the opinion of the Treating Investigator makes the subject unable to complete the study per protocol, e.g.

    * Subject is not likely to avoid other prohibited facial cosmetic treatments;
    * Subject is not likely to complete the study because of other commitments;
    * Subject is anticipated to be unavailable for visits, incapable of understanding the investigational assessments or having unrealistic expectations of treatment result;
    * Subject who has a concomitant condition (e.g. acute viral or bacterial infection with fever) that might confuse or confound study treatments or assessments.
17. Subject who plan to lose or has a medical condition that may cause them to lose a significant amount of weight during the course of the study.
18. Study center personnel, close relatives of the study center personnel (e.g. parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.
19. Participation in any other interventional clinical study within 30 days before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Demonstrate non-inferiority of GP0112 versus a comparator-control in cheek augmentation and correction of midface contour deficiencies | 3 Months
  Investigator's and Blinded Evaluator's live assessment on validated 4-grade photographic Medicis Midface Volume Scale (MMVS) to rate the subject's right and left midface separately for severity of volume deficiency. The change from baseline at Month 3 will be the response variable

SECONDARY OUTCOMES:
Effectiveness of GP0112 and comparator-control based on the validated 4-grade Medicis Midface Volume Scale (MMVS) assessment | 3, 6, 9, 12, 15, 18 and 19 Months
  Responder rate based on the Blinded Evaluator's live assessment of the validated 4-grade Medicis Midface Volume Scale (MMVS). A responder is defined as a subject with at least 1 grade improvement from baseline on both sides of the face concurrently
Effectiveness of GP0112 on the Global Aesthetic Improvement Scale (GAIS) | 3, 6, 9, 12, 15, 18 and 19 Months
  Percentage of responders, defined by having at least "Improved" (improved, much improved or very much improved) on the Global Aesthetic Improvement Scale (GAIS) by the subject and treating investigator
Effectiveness of GP0112 and comparator-control using the FACE-Q | 3, 6, 9, 12, 15, 18 and 19 Months
  Change from baseline in FACE-Q Satisfaction with Cheeks Rasch transformed total score, as well as proportion of subjects in each response category for each of the individual questions for the FACE-Q Satisfaction with Cheeks and Satisfaction with Outcome questionnaires
Effectiveness of GP0112 and comparator-control using Subject Satisfaction Questionnaire (SSQ) | 3, 6, 9, 12, 15,18 and 19 Months
  Proportion of subjects in each response category (strongly agree, agree, neutral, disagree or strongly disagree) for every question in the Subject Satisfaction Questionnaire (SSQ)
Effectiveness of GP0112 and comparator-control in returning to social engagement | 3, 6, 9, 12, 15,18 and 19 Months
  Time in hours until the subject feels comfortable returning to social engagement after treatment, based on subject diary reporting
Safety of GP0112 in cheek augmentation and correction of midface contour deficiencies adverse events (AEs) | Up to 19 Months
  Incidence, intensity, time to onset and duration of adverse events
Safety of GP0112 in cheek augmentation and correction of midface contour pre-defined expected post-treatment events | Up to 19 Months
  Incidence, intensity and number of days of pre-defined expected post-treatment events collected using subject diaries for 28 days following each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (10):
- Canada (10):
  - Galderma Research Site, Calgary, Alberta
  - Galderma Research Site, Edmonton, Alberta
  - Galderma Research Site, Vancouver, British Columbia
  - Galderma Research Site, Winnipeg, Manitoba
  - Galderma Research Site, Oakville, Ontario
  - Galderma Research Site, Richmond Hill, Ontario
  - Galderma Research Site, Toronto, Ontario
  - Galderma Research Site, Windsor, Ontario
  - Galderma Research Site, Woodbridge, Ontario
  - Galderma Research Site, Montreal, Quebec